CLINICAL TRIAL: NCT05800405
Title: A Feasibility Study of Bridging Radiation to All Sites of FDG-Avid Disease for Commercial CAR T-Cell Infusion in Patients With Large B-Cell Lymphoma
Brief Title: Evaluation of Bridging Radiation Therapy Before CAR T-Cell Infusion for the Treatment of Relapsed or Refractory Large B-Cell Lymphoma
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22141; NCI-2023-02190 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 22141 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2023-03-24; First posted 2023-04-05 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Recurrent Diffuse Large B-Cell Lymphoma; Refractory Diffuse Large B-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Specimen Handling; Immunotherapy, Adoptive; Radiation; Leukapheresis; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (leukapheresis, external beam radiation, CAR-T) (Experimental): Patients undergo leukapheresis per standard of care, undergo external beam radiation therapy, and undergo CAR T-cell infusion per standard of care on study. Patients undergo PET/CT throughout the study and may undergo MRI during screening. Patients also undergo blood sample collection throughout the study.
  Interventions: Procedure: Biospecimen Collection; Biological: Chimeric Antigen Receptor T-Cell Therapy; Procedure: Computed Tomography; Radiation: External Beam Radiation Therapy; Procedure: Leukapheresis; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Biological: Chimeric Antigen Receptor T-Cell Therapy — Receive CAR-T per standard of care
  Other Names: CAR T Infusion; CAR T Therapy; CAR T-cell Therapy; Chimeric Antigen Receptor T-cell Infusion
Procedure: Computed Tomography — Undergo PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized Tomography; CT; CT Scan; tomography
Radiation: External Beam Radiation Therapy — Undergo radiation therapy
  Other Names: Definitive Radiation Therapy; EBRT; External Beam Radiation; External Beam Radiotherapy; External Beam RT; external radiation; External Radiation Therapy; external-beam radiation; Radiation, External Beam; Teleradiotherapy; Teletherapy; Teletherapy Radiation
Procedure: Leukapheresis — Receive leukapheresis
  Other Names: Leukocytopheresis; Therapeutic Leukopheresis
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT

SUMMARY:
This early phase I clinical trial evaluates bridging radiation therapy given before chimeric antigen receptor (CAR) T-cell infusion to treat large B-cell lymphoma (LBCL) that has come back (relapsed) or has not responded to previous treatment (refractory). Patients with relapsed or refractory disease have historically poor prognosis. CAR T-cell therapy is a type of treatment in which a patient's T-cells (a type of immune system cell) are changed in the laboratory so they will attack cancer cells. T-cells are taken from a patient's blood (leukapheresis). Then the gene for a special receptor that binds to a certain protein on the patient's cancer cells is added to the T-cells in the laboratory. The special receptor is called a chimeric antigen receptor (CAR). Large numbers of the CAR T-cells are grown in the laboratory and given to the patient by infusion for treatment of certain cancers. While the outcomes from CAR T-cell therapy appear favorable, in the time between leukapheresis and CAR T-cell infusion many patients have symptomatic or life-threatening disease which often requires bridging therapy. Bridging therapy aims to slow disease progression and control symptoms during this critical period prior to CAR T-cell infusion. Radiation therapy uses high energy x-rays, particles, or radioactive seeds to kill cancer cells. Giving bridging radiation therapy to patients with relapsed or refractory LBCL prior to CAR T-cell infusion may improve treatment outcomes with minimal toxicity.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Evaluate if bridging radiation to all sites of F-fluorodeoxyglucose (FDG)-avid disease can be feasibly administered prior to commercial CAR T-cell infusion in patients with large B-cell lymphoma (LBCL).

SECONDARY OBJECTIVES:

I. Assess the toxicities of bridging radiation in patients with LBCL. II. Assess overall response rate, complete response rate, progression-free survival, local control, distant control, and overall survival after bridging radiation and CAR T-cell infusion in patients with LBCL.

EXPLORATORY OBJECTIVES:

I. Bank blood for future immune profiling or other correlatives. II. Explore the association between positron emission tomography (PET)/computed tomography (CT) radiomic features and clinical outcomes.

III. Collect PET/CT imaging data using the RefleXion X1 linear accelerator imaging system.

OUTLINE:

Patients undergo leukapheresis per standard of care, undergo external beam radiation therapy, and undergo CAR T-cell infusion per standard of care on study. Patients undergo PET/CT throughout the study and may undergo magnetic resonance imaging (MRI) during screening. Patients also undergo blood sample collection throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant and/or legally authorized representative.

  * Assent, when appropriate, will be obtained per institutional guidelines.
* Age: >= 18 years.
* Eastern Cooperative Oncology Group (ECOG) =< 2 or Karnofsky Performance Status (KPS) >= 60.
* Histologically confirmed large B-cell lymphoma.
* Relapsed/refractory disease.
* Planned to undergo commercial CAR T-cell infusion within 3 months of enrollment.
* 6 or fewer sites (treatable with a maximum of 3 isocenters) of FDG-PET avid disease, treatable with a a maximum of 3 isocenters.
* Measurable disease e.g., at least 1.5 cm on CT/MRI or by Response Evaluation Criteria in Solid Tumors 1.1 (RECIST 1.1).
* Fully recovered from the acute toxic effects (except alopecia) to =< grade 1 to prior anti-cancer therapy.
* Women of childbearing potential (WOCBP): negative urine or serum pregnancy test (performed within 30 days prior to day 1 of protocol therapy).

  * If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.

Exclusion Criteria:

* Prior CD19-directed therapy.
* Radiation therapy within 21 days prior to day 1 of protocol therapy.
* Central nervous system (CNS) disease.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to study agent.
* Active diarrhea.
* Clinically significant uncontrolled illness.
* Active infection requiring antibiotics.
* Other active malignancy.
* Females only: Pregnant.
* Any other condition that would, in the investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns with clinical study procedures.
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2023-07-20 (Actual); Primary Completion 2027-01-04 (Estimated); Study Completion 2027-01-04 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants completing planned radiation therapy | From the first fraction of radiation until approximately 1 month after infusion of chimeric antigen receptor (CAR) T-cell therapy
  Will be assessed by the proportion of participants completing planned radiation therapy without any grade 3 or higher radiation-attributable (possibly, probably, or definitely) adverse events (AEs), along with its associated 95% Clopper Pearson exact binomial confidence interval (CI). All participants who start protocol radiation therapy are evaluable.

SECONDARY OUTCOMES:
Incidence of AEs | Up to 1 year
  Will be assessed by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version (v)5.0 except in the case of cytokine release syndrome and neurotoxicity, which will be graded by American Society for Transplantation and Cellular Therapy Consensus Grading and not NCI CTCAE v5.0. All participants who receive any fraction of protocol radiation are evaluable.
Objective response rate | Up to 1 year
  Will be defined as the proportion of participants that achieve a best response of either complete response (CR) or partial response after CAR T-cell infusion and prior to disease progression and/or start of other anti-lymphoma therapy, along with its associated 95% Clopper Pearson exact binomial CI. Only participants who receive CAR T-cell infusion post protocol radiation are evaluable.
Complete response rate | Up to 1 year
  Will be defined as the proportion of participants that achieve a best response of CR after CAR T-cell infusion and prior to disease progression and/or start of other anti-lymphoma therapy, along with its associated 95% Clopper Pearson exact binomial CI. Only participants who receive CAR T-cell infusion post protocol radiation are evaluable.
Progression free survival | Time from CAR T-cell infusion to time of disease relapse/progression or death due to any cause, whichever occurs first, assessed up to 1 year
  Will be assessed only in participants who receive CAR T-cell infusion post protocol radiation are evaluable for this endpoint. Will be estimated for patients who received radiation and CAR T-cells using the Kaplan Meier method along with the Greenwood estimator of standard error; 95% confidence interval will be constructed based on log-log transformation.
Overall survival | Time from CAR T-cell infusion to time of death due to any cause, assessed up to 1 year
  Will be assessed only in participants who receive CAR T-cell infusion post protocol radiation are evaluable. Will be estimated for patients who received radiation and CAR T-cells using the Kaplan Meier method along with the Greenwood estimator of standard error; 95% confidence interval will be constructed based on log-log transformation.
Local control | Time from CAR T-cell infusion to time of disease relapse/progression within the radiation field, assessed up to 1 year
  Will be defined as the 80% isodose line. Only participants who receive CAR T-cell infusion post protocol radiation are evaluable. Will be analyzed by competing risk method where death without any progression will also be treated as a competing risk event.
Distant control | Time from CAR T-cell infusion to time of disease relapse/progression outside the radiation field, assessed up to 1 year
  Will be defined as the 80% isodose line. Only participants who receive CAR T-cell infusion post protocol radiation are evaluable. Will be analyzed by competing risk method where death without any progression will also be treated as a competing risk event.

CONTACTS AND LOCATIONS:
Overall Officials: Savita V Dandapani, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States